CLINICAL TRIAL: NCT03484663
Title: Small Catheter Drainage With Chest Tube After Uniport Video-assisted Thoracoscopic Procedures
Brief Title: Small Catheter Drainage With Chest Tube Versus Chest Tube Alone After Uniport Video-assisted Thoracoscopic Procedures
Acronym: uniportal VATS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, ali mohamed abdelraouf, Doctor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: uniport VATS
Record Dates: First submitted 2018-03-14; First posted 2018-04-02 (Actual); Last update posted 2018-06-11 (Actual); Status verified 2018-06

CONDITIONS: Lung Diseases
MeSH Terms: conditions — Lung Diseases | interventions — Central Venous Catheters

STUDY DESIGN:
Intervention Model Description: case of small catheter drainage with chest tube versus chest tube alone after uniport vats
Who Masked: Participant
Masking Description: patient who will do vats procedure
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Small catheter with chest tube after uniport vats (Experimental): Insertion of small catheter drainage in the same opening with chest tube after uniport vats
  Interventions: Device: central venous catheter (small catheter drainage)
- Chest tube only after uniport vats (No Intervention): After uniport vats we put chest tube only

INTERVENTIONS:
Device: central venous catheter (small catheter drainage) — Insertion central venous catheter ( small catheter drainage ) after uniport vats to decrease hospital stay and to easy drainage after procedure
  Arms: Small catheter with chest tube after uniport vats

SUMMARY:
Small catheter drainage with chest tube after uniport Video-assisted Thoracoscopic Procedures

DETAILED DESCRIPTION:
Traditionally an Intercostal Tube is applied intraoperative following VATS procedures to drain the remaining pneumothorax and residual effusion , some of the residual effusion can't drain by intercostal tube which lead to prolonged hospital stay hypothesis that putting an additional small catheter drainage at the most depended part of hemithoracic early removal of chest tube without add more pain or hospital stay to the patient.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing uniport video-assisted thoracoscopic surgery at Assiut University Hospital who need intercostal drainage postoperative

Exclusion Criteria:

* Patients who do not need intercostal tube post operative

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2018-10-01 (Estimated); Primary Completion 2019-05-01 (Estimated); Study Completion 2019-07-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with failure of initial intervention | one year
  Number of participants with failure of initial intervention , Requiring a second intervention i.e.insert second tube